CLINICAL TRIAL: NCT05134896
Title: Visual Performance After Optically Correcting the Eye's Aberration With a Spatial Light Modulator
Brief Title: Visual Performance With Spatial Light Modulator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Geunyoung Yoon, Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00003209
Record Dates: First submitted 2021-11-11; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Normal Healthy Eyes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- normal healthy group (Experimental): Spatial light modulator
  Interventions: Device: Spatial light modulator

INTERVENTIONS:
Device: Spatial light modulator — This device compensates for the eye's optical imperfections (aberrations) at the foveal and peripheral retina.

SUMMARY:
Eye's aberrations have been known to degrade human visual performance and the visual performance is significantly improved when correcting the aberrations in the central visual field. However, how the aberration correction affects the peripheral visual performance is not well understood. Moreover, how central and peripheral vision interacts remains unclear.

To conduct the study, we will use an adaptive optics vision simulator equipped with a Shack-Hartmann wavefront sensor and a spatial light modulator (see details in procedures section of the protocol). This system is capable of noninvasively controlling the eye's optical quality and evaluating visual performance simultaneously over a wide area of visual space. This study provides insights into the visual performance in the periphery visual field, and interaction between central and peripheral visual fields.

The goal of this study is to evaluate the visual performance at central and peripheral visual fields after correcting the ocular aberrations. An optical system equipped with a liquid crystal spatial light modulator will be used to achieve this goal non-invasively.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

* Is between the ages of 18 and 60.
* Has normal corneas i.e. no corneal infections, no systemic pink eye, no clinically significant dry eye, and no corneal dystrophies.
* Has refractive errors less than +/- 10.0 Diopters in both eyes.

Exclusion Criteria:

A person will be excluded from the study if he/she:

* Adults between the ages of 18-60 who are unable to give informed consent
* Individuals below 18 years old
* Individuals above the age of 60
* Pregnant women (self-reporting, hormonal changes may alter the refractive status of the eye)
* Prisoners
* Students for whom you have direct access to/influence on grades
* People who do not understand or speak English
* Has clinically significant dry eye.
* Has clinically significant cataract.
* Has spherical refractive error that exceeds the limits outlined above.
* Is unable to hold his or her head steady for the duration of study measurements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | up to 6 separate sessions (each session taking up to 2 hours)
  Snellen "Tumbling E" method will be used to determine the smallest letter that a subject can see.
Contrast sensitivity | up to 6 separate sessions (each session taking up to 2 hours)
  Light and dark sinusoidal stripes (Gabor gratings) will used to determine the smallest contrast that a subject can see
Contrast perception | up to 6 separate sessions (each session taking up to 2 hours)
  Light and dark sinusoidal stripes (Gabor gratings) will used to determine differences in contrast perceived by the central and peripheral visual system

IPD SHARING:
Plan to Share IPD: No